CLINICAL TRIAL: NCT03684967
Title: An Open-label Single Arm Multi-center Phase II Study to Assess Fruquintinib in High Risk Patients With Advanced Non-squamous Non-small Cell Lung Cancer
Brief Title: Study of Fruquintinib (HMPL-013) in High Risk Patients With Advanced NSCLC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the study stopped because the company's strategy.
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-013-00CH2
Record Dates: First submitted 2018-08-23; First posted 2018-09-26 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2018-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fruquintinib (Experimental): Fruquintinib treatment: administration for 3 weeks followed by 1 week break, and administration every day for the first 21 days.
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib treatment: 4mg in the Cycle 1,administration for 3 weeks followed by 1 week break, and administration every day for the first 21 days.5mg ,administration for 3 weeks followed by 1 week break, and administration every day for the first 21 days

SUMMARY:
Fruquintinib administered at 4 mg once daily in cycle 1 and 5 mg once daily in followed cycles (3 weeks on and 1 week off, 4 weeks as 1 cycle) was well tolerated and demonstrated encouraging preliminary clinical antitumor activity in patients with advanced NSCLC in phase II study.

This study is aimed to evaluate the efficacy and safety of Fruquintinib in the treatment of high risk patients with advanced NSCLC who is > 75 years, or Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) = 2, or without systemic chemotherapy, or with at least three lines systemic chemotherapies.

DETAILED DESCRIPTION:
This is an open-label single arm multi-center phase II study to assess the efficacy and safety of Fruquintinib in high risk patients with advanced NSCLC who is > 75 years, or ECOG PS = 2, or without systemic chemotherapy, or with at least three lines systemic chemotherapies.

After checking eligibility criteria, subjects will take Fruquintinib as below: 4 mg once daily in the Cycle 1, administration for 3 weeks followed by 1 week break. 5mg once daily in followed cycles, administration for 3 weeks followed by 1 week break.

Primary Efficacy Endpoint:

Disease Control Rate (DCR) (According to RECIST Version 1.1). Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

Secondary Efficacy Endpoints:

Objective Response Rate (ORR), Duration of Response (DOR), Progression free survival (PFS), Overall Survival (OS) and Quality of Life (QoL).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Histologically or cytological documented stage IIIB/IV non-squamous non-small cell lung cancer patients
* Epidermal growth factor receptor (EGFR) mutation wild type; or EGFR activating mutation and resistant / intolerant to related targeted therapies
* Anaplastic lymphoma kinase (ALK) mutation negative; or ALK mutation positive and resistant / intolerant to related targeted therapies
* Presence of at least one measurable tumor lesion in accordance with RECIST 1.1 criteria
* Expected survival > 12 weeks
* Queue 1: 1) Age > 75 years 2) Disease progression during or within 3 months after first-line systemic chemotherapy; or intolerable toxicity / intolerance during first-line systemic chemotherapy (excluding immunotherapy); or without systemic chemotherapy (rejected or intolerable), judged by investigators 3) Eastern Cooperative Oncology Group (ECOG) of 0-1
* Queue 2: 1) Age 18-75 years old (including 18 and 75 years old) 2) Disease progression during or within 3 months after first-line systemic chemotherapy; or intolerable toxicity / intolerance during first-line systemic chemotherapy (excluding immunotherapy); or without systemic chemotherapy (rejected or intolerable), judged by investigators 3) Eastern Cooperative Oncology Group (ECOG) of 2
* Queue 3: 1) Age 18-75 years old (including 18 and 75 years old) 2) without systemic chemotherapy 3) Eastern Cooperative Oncology Group (ECOG) of 0-1
* Queue 4: 1) Age 18-75 years old (including 18 and 75 years old) 2) Disease progression during or within 3 months after at least three lines systemic chemotherapy; or intolerable toxicity / intolerance during at least third-line systemic chemotherapy (excluding immunotherapy) 3) Eastern Cooperative Oncology Group (ECOG) of 0-1

Exclusion Criteria:

* Patients who have participated in another clinical trial or received systemic anti-neoplastic chemotherapy, biotherapy or immunotherapy within 3 weeks prior to administration of the study drug; or received target drugs treatment as EGFR - Tyrosine Kinase Inhibitors (TKIs), ALK inhibitors, within in 2 weeks; or received anti-neoplastic traditional Chinese medicine within 1 week; or received pleural infusion chemotherapy within 1 week.
* Patients who have received palliative radiotherapy within 1 week prior to administration of the study drug; or received radical / extensive radiotherapy within 3 weeks; or received brachytherapy within 60 days (as seed implantation)
* Patients who have previously received therapy with VEGFR inhibitors
* Patients who have previously received potent inhibitor and/or potent inducer of cytochrome P450 3A4 (CYP3A4) within two 2 weeks prior to administration of the study drug; receiving P-glycoprotein (P-gp) and breast cancer resistance protein (BCRP) substrate drugs within two 2 weeks prior to randomization
* Patients who have previously received major surgery or large invasive procedure within 60 days prior to administration of the study drug, or incomplete recovery from previous surgery/procedure, or incomplete healing of surgical incision/wound; no recovery of the toxicity from previous antitumor therapies (i.e., CTCAE grade > 1) (if applicable)
* Patients with brain metastasis
* Patients with spinal compression with no surgical therapy and/or radical radiotherapy; or previously treated spinal compression, however, no clinical evidence showing stable condition
* Radiological evidence showing tumor invading or encompassing major blood vessels of lungs (e.g., pulmonary artery, superior vena cava)
* Patients with other primary malignancies within the past 5 years except basal cell carcinoma of skin or carcinoma in situ of cervix
* Patients with uncontrolled active infections, e.g. acute pneumonia
* Patients with active hepatitis B or active hepatitis C, etc. (for patients with a history of hepatitis B, whether treated or not, hepatitis B virus (HBV) DNA ≥500copies or ≥ 100IU / ml)
* Patients with human immunodeficiency virus (HIV) infection
* Patients with dysphagia or known drug malabsorption
* Patients active duodenal ulcer, ulcerative colitis, intestinal obstruction and other gastrointestinal diseases or other conditions that may lead to gastrointestinal bleeding or perforation according to the investigators' judgment; or with a history of intestinal perforation or intestinal fistula
* Patients fulfilling any of the following criteria shall be excluded:

  1. Absolute neutrophil count (ANC) <1.5×109/L, platelet <100×109/L or hemoglobin <9 g/dL within 2 week prior to administration of the study drug
  2. Serum total bilirubin > 1.5 × upper limit of normal (ULN), alanine transaminase and aspartate aminotransferase >2.5×ULN (according to reference range in each clinical study site); ALT and AST > 5×ULN in patients with liver metastasis
  3. Clinically significant electrolyte abnormality
  4. Blood creatinine > ULN and creatinine clearance <50 ml/min
  5. Urine protein 2+ or more, or urine protein quantification ≥1.0 g/24 h
  6. Activated partial thromboplastin time (APTT) or/and INR and prothrombin time (PT) > 1.5×ULN (according to reference range in each clinical study site)
* Patients with uncontrolled hypertension, systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg after symptomatic treatment
* Cardiac function: left ventricular ejection fraction <50% (by echocardiography); moderate or above mitral or tricuspid insufficiency; acute myocardial infarction, serious/unstable angina pectoris or coronary artery bypass grafting within 6 months prior to randomization; or New York heart association (NYHA) grade 2 or above cardiac insufficiency
* Patients who have a history of arterial thrombosis or deep venous thrombosis within 6 months prior to administration of the study drug; history or evidence of thrombosis or bleeding tendency regardless of the severity within 2 months; history of hemoptysis (i.e. coughing blood in bright red color at least 2.5ml or 1/2 teaspoon) within 2 weeks; history of liver hemangioma > 3 cm
* Patients who have a history of stroke and/or transient ischemic attack within 12 months prior to administration of the study drug
* Patients with skin wound, surgical site, wound site, severe mucosal ulcer or fracture without complete healing
* Pregnant or lactating women, or women of child bearing potential with positive pregnancy test result before the first dose; Patients with child bearing potential who or whose sexual partners are not willing to take contraceptive measures
* Patients with any clinical or laboratory abnormalities unsuitable for participating in this clinical trial according to the investigator's judgment
* Patients with serious psychological or psychiatric disorders which may affect subject compliance in this clinical study
* Patients who are allergic to analogue of Fruquintinib and/or its inactive ingredients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | from the first dose until progressive disease or End of Therapy (EOT) due to any cause, whichever came first, assessed up to 8 weeks.
  Tumor assessment will be performed using radiography method at the first 4th week and 8th week after the first dose, or until the occurrence of progressive disease (PD), using RECIST v 1.1.
Safety and tolerance evaluated by incidence, severity and outcomes of AEs | from the first dose to 30 days post the last dose
  Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 4.03

SECONDARY OUTCOMES:
Objective response rate (ORR) | from the first dose until progressive disease or EOT due to any cause, whichever came first, assessed up to 1 year
  Tumor assessment will be performed using radiography method at the first 4th week and 8th week after the first dose, then every 8 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1.
Duration of Response (DOR) | from the first dose until progressive disease or EOT due to any cause, whichever came first, assessed up to 1 year
  Tumor assessment will be performed using radiography method at the first 4th week and 8th week after the first dose, then every 8 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1.
Progression free survival (PFS) | from the first dose until progressive disease or EOT due to any cause, whichever came first, assessed up to 1 year
  Tumor assessment will be performed using radiography method at the first 4th week and 8th week after the first dose, then every 8 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1.
Overall survival (OS) | from the first dose until death due to any cause, assessed up to 3 year
  Every two months follow up after EOT observation period at 30 days after the last medication
Quality of Life (QoL) | from the first dose to 30 days post the last dose
  The change of QoL will be assessed by the EORTC Quality of Life Questionnaire Core-30 (QLQ-C30) plus QLQ-Lung Cancer 13-item (LC13) ( LC13 is a supplementary module plus QLQ-C30 as one complete measure) every 4 weeks. A descriptive statistics analysis will be used to look at QoL over the time course.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China